CLINICAL TRIAL: NCT00000491
Title: Aspirin-Myocardial Infarction Study (AMIS)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Prevention
Other Study IDs: 10
Record Dates: First submitted 1999-10-27; First posted 1999-10-28 (Estimated); Last update posted 2016-03-25 (Estimated); Status verified 2012-04

CONDITIONS: Cardiovascular Diseases; Coronary Disease; Heart Diseases; Myocardial Infarction; Myocardial Ischemia
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Disease; Heart Diseases; Myocardial Infarction; Myocardial Ischemia | interventions — Aspirin

INTERVENTIONS:
Drug: aspirin

SUMMARY:
To determine whether the daily administration of 1 gm of aspirin to individuals with a documented myocardial infarction would result in a significant reduction in mortality over a three year period.

DETAILED DESCRIPTION:
BACKGROUND:

It had been postulated that thrombosis plays a major role in the late stages of coronary artery occlusion. Platelet aggregation is a large component in the formation of arterial thrombi. Theoretically, an agent which prevents the aggregation of platelets would be of value in people with coronary artery disease. Aspirin, in small doses, inhibits platelet aggregation for prolonged periods of time, and therefore might be expected to prevent or retard the occlusion of coronary arteries. This would be reflected in a decrease in the incidence of myocardial infarction and a decrease in mortality due to coronary artery disease.

Several studies had given preliminary evidence that regular administration of aspirin may be of benefit to patients with known coronary artery disease. A National Heart and Lung Institute-sponsored study, the Coronary Drug Project, ran a pilot trial of aspirin and placebo in men with previous myocardial infarctions. Preliminary results from this trial demonstrated its feasibility and led NHLBI to sponsor a more definitive controlled study of the benefit of aspirin in the secondary prevention of coronary heart disease.

An Institute Planning Committee met four times between October 1974 and April 1975 and developed a protocol, manual of operations, and data collection forms. Recruitment of patients began in June 1975, with the first patient randomized on July 2, 1975. Patients who were randomized had been seen at the AMIS Clinical Center for two initial visits and one baseline visit and were free of any reasons for exclusion, such as the current use of anticoagulants and a history of adverse reactions to aspirin. Patients took acetaminophen at times when they would normally take aspirin.

Follow-up was for a minimum of 3 years, with each patient seen at 4-month intervals and monitored for side effects and various nonfatal events, including cardiovascular problems. The primary endpoint was mortality. Annually, a detailed history was obtained and a complete physical examination performed. The study involved 30 clinical centers, a coordinating center, and a central laboratory.

The study completed patient recruitment in the scheduled one year period. A total of 4,524 post-MI patients were enrolled by the 30 clinical centers. Three-year minimum patient follow-up ended in August 1979.

DESIGN NARRATIVE:

Randomized, double-blind, fixed sample. Eligible patients were assigned to a treatment group receiving 1 gm of aspirin daily (the equivalent of three standard aspirin tablets) or to a control group receiving a placebo.

ELIGIBILITY:
Men and women, ages 30 to 69. Had a documented myocardial infarction.

Ages: 30 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1974-10; Study Completion 1979-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Allan Barker — Salt Lake Clinic Research Foundation; David Berkson — Unity Health Toronto; William Berstein — Icahn School of Medicine at Mount Sinai; Nemat Borhani — University of California, Davis; Elmer Cooper — Santa Rosa Medical Center; Leonard Dreifus — Lankenau Hospital; Noble Fowler — University of Cincinnati; Phillip Frost — USPHS Hospital; Mario Garcia-Palmieri — University of Puerto Rico Medical Science Campus; Hugh Gilmore — University of Miami; Sidney Goldstein — Henry Ford Hospital; Olga Haring — Northwestern University; J. Hoover — University of Washington; Richard Hutchinson — University of Mississippi Medical Center; William Krol — University of Maryland at Baltimore; Peter Kuo — Rutgers Medical School; Charles, Laubach — Institute for Medical Education and Research; Bernard Lewis — Palo Alto Medical Research Foundation; Jessie Marmorston — University of Southern California; J. McNamara — Pacific Health Research Institute; Dayton Miller — U.S. Centers for Disease Control and Prevention; Thaddeus Prout — Greater Baltimore Medical Center; David Richardson — Virginia Commonwealth University; Jorge Rios — George Washington University; Paul Samuel — Long Island Jewish-Hillside Medical Center; Stephen Scheidt — Weill Medical College of Cornell University; Robert Schlant — Emory University; Henry Schoch — University of Michigan; James Schoenberger — Rush University Medical Center; Marvin Segal — MOUNT SINAI HOSPITAL; Pantel Vokonas — Boston Health and Hospitals Department; C. Williams — Ogden Research Foundation; Gary Wilner — Endeavor Health

REFERENCES:
- [Background] Aspirin Myocardial Infarction Research Group: A Study of Aspirin in Patients with Myocardial Infarction. Prostaglandins in Hematology. Spectrum Publications Inc, New York, l977, 36l-370.
- [Background] An intervention study-the aspirin myocardial infarction study. Lipids. 1977 Jan;12(1):59-63. doi: 10.1007/BF02532973. PMID 319319
- [Background] A randomized, controlled trial of aspirin in persons recovered from myocardial infarction. JAMA. 1980 Feb 15;243(7):661-9. PMID 6985998
- [Background] Aspirin Myocardial Infarction Research Group: Aspirin Myocardial Infarction Study: Design, Methods and Baseline Results. DHEW Pub. No. (NIH) 80-2l06, l980.
- [Background] The aspirin myocardial infarction study: final results. The Aspirin Myocardial Infarction Study research group. Circulation. 1980 Dec;62(6 Pt 2):V79-84. PMID 7438383
- [Background] Wasserman AG, Bren GB, Ross AM, Richardson DW, Hutchinson RG, Rios JC. Prognostic implications of diagnostic Q waves after myocardial infarction. Circulation. 1982 Jun;65(7):1451-5. doi: 10.1161/01.cir.65.7.1451. PMID 7042113
- [Background] Goldstein S, Friedman L, Hutchinson R, Canner P, Romhilt D, Schlant R, Sobrino R, Verter J, Wasserman A. Timing, mechanism and clinical setting of witnessed deaths in postmyocardial infarction patients. J Am Coll Cardiol. 1984 May;3(5):1111-7. doi: 10.1016/s0735-1097(84)80167-9. PMID 6423716
- [Background] Mattson ME, Curb JD, McArdle R. Participation in a clinical trial: the patients' point of view. Control Clin Trials. 1985 Jun;6(2):156-67. doi: 10.1016/0197-2456(85)90121-7. PMID 4006489
- [Background] Shekelle RB, Gale M, Norusis M. Type A score (Jenkins Activity Survey) and risk of recurrent coronary heart disease in the aspirin myocardial infarction study. Am J Cardiol. 1985 Aug 1;56(4):221-5. doi: 10.1016/0002-9149(85)90838-0. PMID 3895879
- [Background] Frost PH, Verter J, Miller D. Serum lipids and lipoproteins after myocardial infarction: associations with cardiovascular mortality and experience in the Aspirin Myocardial Infarction Study. Am Heart J. 1987 Jun;113(6):1356-64. doi: 10.1016/0002-8703(87)90648-x. PMID 3591604
- [Background] Schoenberger JA. Recruitment experience in the Aspirin Myocardial Infarction Study. Control Clin Trials. 1987 Dec;8(4 Suppl):74S-78S. doi: 10.1016/0197-2456(87)90009-2. PMID 3440392
- [Background] Furberg CD, Friedman LM, MacMahon SW: Women as Participants in Trials of the Primary and Secondary Prevention of Cardiovascular Disease: Part II. Secondary Prevention: The Beta-Blocker Heart Attack Trial and the Aspirin Myocardial Infarction Study, in: Coronary Heart Disease in Women. ED Eaker, B Packard, NK Wenger, TB Carkson, HA Tyroler (Eds). New York, Haymarket Doyma, pp 241-246, 1987.
- [Background] Howard J, Whittemore AS, Hoover JJ, Panos M. How blind was the patient blind in AMIS? Clin Pharmacol Ther. 1982 Nov;32(5):543-53. doi: 10.1038/clpt.1982.201. PMID 7127995
- Available data/document: Individual Participant Data Set: AMIS — http://biolincc.nhlbi.nih.gov/studies/amis/ — NHLBI provides controlled access to IPD through BioLINCC. Access requires registration, evidence of local IRB approval or certification of exemption from IRB review, and completion of a data use agreement.